CLINICAL TRIAL: NCT00554307
Title: Comparison of Cerebral, Renal and Mesenteric Perfusion Using Near Infrared Spectroscopy in Neonates During Patent Ductus Arteriosus Closure With Ibuprofen or Indomethacin.
Brief Title: Brain, Gut and Kidney Blood Flow During Medical Closure of PDA
Status: Withdrawn | Type: Observational
Why Stopped: Not able to enroll patients
Sponsor: University of Louisville (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: DStewart, ULouisville
Other Study IDs: UofL IRB 328.07
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Patent Ductus Arteriosus
Keywords: patent ductus arteriosus; indomethacin; neoprofen; blood flow
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Indo: Infants that are treated with indomethacin
  Interventions: Device: INVOS Cerebral/Somatic oximeter
- Neo: Infants treated with neoprofen
  Interventions: Device: INVOS Cerebral/Somatic oximeter
- Control: Infants without PDA
  Interventions: Device: INVOS Cerebral/Somatic oximeter

INTERVENTIONS:
Device: INVOS Cerebral/Somatic oximeter — Placement of sensors on back, abdomen and forehead for measurement of perfusion beginning 1 hour prior to initiation of drug, during medical treatment for PDA and for 24 hours after the last dose. For control infants, monitoring will continue for 48 hours.

SUMMARY:
The purpose of this study is to determine how the medications which are used to close the patent ductus arteriosus (PDA) in preterm infants affect brain, kidney and gut blood flow when compared to infants that are not treated with these medications. The medications being used for PDA closure are indomethacin and neoprofen.

DETAILED DESCRIPTION:
All babies requiring medical treatment of their PDA will receive up to 3 doses of medication. For babies enrolled in the control group of this study, she/he will not be treated with either of these medicines.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 32 weeks gestation;
* Less than or equal to 1250 g;
* Mechanical ventilation;
* Echocardiographic findings of PDA with left to right shunting;
* Medical judgement of neonatologist for medical treatment;

Exclusion Criteria:

* Urine output less than 1 ml/k/hr over previous 12 hours;
* Serum creatinine greater than 1.5 mg/dL;
* Platelet count less than 100,000 per cubic mm;
* Significant skin breakdown at sensor areas;
* Significant congenital anomalies
* Intraventricular hemorrhage greater than or equal to grade III

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants with patent ductus arteriosus requiring medical intervention
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Changes in blood flow from baseline in infants treated with indomethacin or neoprofen. Blood flow will be measured in the brain, kidney and mesentery. | 48-72 hours
Measure oxygenation/blood flow to brain during PDA treatment | Study period

SECONDARY OUTCOMES:
Oxygenation during/after treatment with PDA therapy | Study period

CONTACTS AND LOCATIONS:
Overall Officials: Dan L Stewart, MD, Principal Investigator — University of Louisville
Locations (1):
- Kosair Children's Hospital, Lousiville, Kentucky, United States